CLINICAL TRIAL: NCT06652763
Title: Manganese-enhanced Magnetic Resonance Imaging (MEMRI) in Heart Failure With Preserved Ejection Fraction
Acronym: MEMRI in HFpEF
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0883
Record Dates: First submitted 2023-11-27; First posted 2024-10-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Echocardiography; Walk Test; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma will be stored for future analyses including established biomarkers and discovery studies such as proteomic, lipidomic, metabolomic and genomic analyses and other new methodologies that may be developed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- HFpEF with T2D: Participants with heart failure with preserved ejection fraction and type 2 diabetes
  Interventions: Other: Minnesota Living with Heart Failure Questionnaire; Diagnostic Test: Echocardiogram; Diagnostic Test: Six-minute walk test; Diagnostic Test: Manganese-enhanced MRI and 31-P magnetic resonance spectroscopy; Diagnostic Test: Cardiovascular magnetic resonance scan; Diagnostic Test: Blood tests
- HFpEF without T2D: Participants with heart failure with preserved ejection fraction but without type 2 diabetes
  Interventions: Other: Minnesota Living with Heart Failure Questionnaire; Diagnostic Test: Echocardiogram; Diagnostic Test: Six-minute walk test; Diagnostic Test: Manganese-enhanced MRI and 31-P magnetic resonance spectroscopy; Diagnostic Test: Cardiovascular magnetic resonance scan; Diagnostic Test: Blood tests
- Controls: Healthy volunteers without heart failure or type 2 diabetes
  Interventions: Other: Minnesota Living with Heart Failure Questionnaire; Diagnostic Test: Echocardiogram; Diagnostic Test: Six-minute walk test; Diagnostic Test: Manganese-enhanced MRI and 31-P magnetic resonance spectroscopy; Diagnostic Test: Cardiovascular magnetic resonance scan; Diagnostic Test: Blood tests

INTERVENTIONS:
Other: Minnesota Living with Heart Failure Questionnaire — Self-administered, validated questionnaire to assess symptoms of heart failure
Diagnostic Test: Echocardiogram — Resting transthoracic echocardiogram to exclude valvular pathology and the assess indices of systolic and diastolic function and speckle tracking for strain
Diagnostic Test: Six-minute walk test — Standardised, objective assessment of exercise capacity
Diagnostic Test: Manganese-enhanced MRI and 31-P magnetic resonance spectroscopy — Using a 3-Tesla scanner, 31P magnetic resonance spectroscopy will be performed to obtain information regarding cardiac energetics. An intravenous infusion of manganese dipyridoxyl diphosphate (mangafodipir, MnDPDP) will be commenced at a rate of 1mL/min using a dose of 5µmol/kg (0.1mL/kg).
Diagnostic Test: Cardiovascular magnetic resonance scan — Scan including adenosine stress perfusion
Diagnostic Test: Blood tests — Full blood count, Urea and electrolytes, Liver function tests, Glucose and HbA1c, Insulin and C-peptide, NTproBNP, High sensitive troponin I, storage of plasma for future analyses

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a condition in which the heart cannot fill with blood effectively. As a result, people with HFpEF suffer fatigue, breathlessness, and develop swollen limbs. The condition often requires multiple admissions to hospital and is associated with a marked loss of lifespan.

Despite being so common, very little is known about why people develop HFpEF and there are hardly any known treatments. Type 2 diabetes (T2D) is a major risk factor for HFpEF, and people with both HFpEF and diabetes are at a heightened risk of hospitalisation and premature death. It is unclear why the combination of diabetes and HFpEF is particularly harmful. This may be related to the hearts of people with type 2 diabetes being unable to take up the mineral calcium properly, as well as due to their hearts being less energy efficient. Both of these are vital to heart muscle pumping and filling, but until recently it has not been possible to assess these in humans.

New advances in heart MRI scans, with dedicated scanner techniques and dyes (manganese contrast), now allow extremely detailed pictures of heart structure, function, calcium uptake and energy efficiency, all during the same scan. The investigators will enlist 40 volunteers with HFpEF (20 with T2D and 20 without T2D), and up to 20 healthy volunteers, to undergo a heart MRI scan with manganese contrast to assess calcium uptake and energy efficiency. This will allow the comparison of people with HFpEF with and without T2D, to see how their hearts are different to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent
* Symptoms (e.g. breathlessness, orthopnoea, ankle swelling, fatigue), signs (e.g. elevated jugular venous pressure, peripheral oedema, third heart sound) or established diagnosis of HF with LV ejection fraction ≥ 50%, or
* Meets HFpEF diagnostic criteria in accordance with the HFA-PEFF diagnostic algorithm form the Heart Failure Association of the European Society of Cardiology, in which a score ≥5 points confirms diagnosis of HFpEF

Exclusion Criteria:

* Known diagnosis of Type 1 Diabetes
* Pregnancy or breast-feeding or females of child bearing age without a negative pregnancy test
* Receiving an investigational drug or device within 30 days prior to participating in the study
* Decompensated heart failure or pulmonary oedema
* History of prolonged corrected QT interval or torsades de pointes
* Second- or third-degree atrioventricular block
* Abnormal liver function tests (> 3x upper limit of normal) or history of liver disease
* Baseline eGFR < 30mL/min/1.73m2
* Any contraindications to MRI including implanted devices/pacemakers
* Severe native valve disease, restrictive cardiomyopathy, constrictive pericarditis or hypertrophic cardiomyopathy, myocarditis or takotsubo cardiomyopathy.
* Recent myocardial infarction within the previous 3 months
* Known diagnosis of pheochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary and secondary care patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Ki | Baseline
  Manganese influx constant as measured by MEMRI scan

SECONDARY OUTCOMES:
T1 values | Baseline
  T1 values measured at 30 minutes post contrast on MEMRI scan
Myocardial PCr/ATP ratio | Baseline
  Phosphocreatine-to-ATP ratio as measured by 31P-magnetic resonance spectroscopy
Left ventricular ejection fraction | Baseline
  %, measured by CMR
LV global longitudinal strain | Baseline
  %, measured by CMR
LV global circumferential strain | Baseline
  %, measured by CMR
LV PEDSR | Baseline
  1/s, measured by CMR
LV mass | Baseline
  grams, measured by CMR
LV mass/volume ratio | Baseline
  Measured by CMR
Myocardial fibrosis | Baseline
  CMR assessed markers of LV myocardial fibrosis (extracellular volume)
Myocardial Perfusion | Baseline
  CMR assessed markers of perfusion (myocardial perfusion reserve)
Associations of Ki with resting PCr/ATP | Baseline
  Univariate and multivariate models to look for association between Ki and PCr/ATP ratio
Associations of exercise capacity with Ki and PCr/ATP in HFpEF | Baseline
  Ki values as assessed by MEMRI, myocardial PCr/ATP as measured by 31P-MRS and six minute walk test distance. Associations will be assessed using univariate and multivariate models.
Plasma biomarkers of metabolic dysregulation, fibrosis and inflammation | Baseline
  This exploratory outcome will assess the differences in a wide range of plasma biomarkers between groups and their association with Ki
10-year outcomes | Baseline
  10-year outcomes including HF hospitalisation (time to first event and cumulative) and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Gerry P McCann, MD, Principal Investigator — University of Leicester; Abhishek Dattani, MBBS, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom